CLINICAL TRIAL: NCT07064980
Title: Analysis of the Effectiveness and Safety of Endoscopic Retrograde Cholangiopancreatography Versus Percutaneous Transhepatic Biliary Drainage in Severe Acute Cholangitis Caused by Common Bile Duct Stones
Brief Title: ERCP Versus PTBD for Severe Acute Cholangitis Caused by Bile Duct Stones
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wuhan Integrated Traditional Chinese and Western Medicine Hospital (Other)
Responsible Party: Principal Investigator, Liping Zhu, Principal Investigator, Wuhan Integrated Traditional Chinese and Western Medicine Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-2021-KY027
Record Dates: First submitted 2025-07-01; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Severe Acute Cholangitis
Keywords: Endoscopic retrograde cholangiopancreatography; Percutaneous transhepatic biliary drainage; Severe Acute Cholangitis; Common Bile Duct Stones
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (ERCP) (Experimental): Patients assigned to this arm underwent endoscopic retrograde cholangiopancreatography (ERCP). After intravenous anesthesia, a duodenoscope was advanced to the major duodenal papilla. The bile duct was cannulated, and common bile duct stones were extracted using a basket or balloon, typically following a biliary sphincterotomy. A nasobiliary tube was placed for drainage. All patients in this group received prophylactic rectal indomethacin (100mg).
  Interventions: Procedure: Endoscopic Retrograde Cholangiopancreatography
- Active Comparator Group (PTBD) (Active Comparator): Patients assigned to this arm underwent percutaneous transhepatic biliary drainage (PTBD). Under general anesthesia and ultrasound guidance, a dilated intrahepatic bile duct was punctured. A guidewire was passed into the biliary system, followed by the placement of an 8-10 Fr drainage catheter for either internal-external or purely external biliary drainage.
  Interventions: Procedure: Percutaneous Transhepatic Biliary Drainage

INTERVENTIONS:
Procedure: Endoscopic Retrograde Cholangiopancreatography — Performed under intravenous anesthesia. A duodenoscope was advanced to the major duodenal papilla. After cannulation and cholangiography, purulent bile was aspirated. Biliary sphincterotomy was performed in most patients (95.2%), followed by stone extraction using a balloon catheter or basket. A 7-10 Fr nasobiliary tube was placed for drainage in all patients. Prophylactic rectal indomethacin (100mg) was also administered.
  Arms: Experimental Group (ERCP)
Procedure: Percutaneous Transhepatic Biliary Drainage — Performed under general anesthesia with endotracheal intubation and ultrasound guidance. An 18G needle was used to puncture a dilated intrahepatic bile duct. After guidewire placement, an 8-10 Fr drainage catheter was inserted for either internal-external drainage (if the guidewire could pass into the duodenum) or purely external biliary drainage.
  Arms: Active Comparator Group (PTBD)

SUMMARY:
This study is a prospective, randomized controlled trial designed to compare the effectiveness and safety of endoscopic retrograde cholangiopancreatography (ERCP) with percutaneous transhepatic biliary drainage (PTBD) for the treatment of severe acute cholangitis caused by common bile duct stones. The primary goal is to determine which emergency drainage procedure leads to faster patient recovery, specifically by evaluating the length of hospital stay, without increasing complication rates.

DETAILED DESCRIPTION:
Severe acute cholangitis (AC) due to common bile duct stones is a life-threatening condition requiring urgent biliary decompression. While both ERCP and PTBD are established minimally invasive options, the optimal choice remains under discussion. This single-center, prospective, randomized controlled trial was conducted to compare these two interventions. A total of 126 patients with severe AC (Tokyo Guidelines 2018 Grade II or III) were randomized to either the ERCP group (n=63) or the PTBD group (n=63). Randomization was performed using a computer-generated sequence with concealed allocation. While operators could not be blinded, outcome assessors and data analysts were. The study hypothesis is that ERCP, as a more direct route for potential stone removal and drainage, may facilitate a quicker overall recovery compared to PTBD. The trial evaluates procedural outcomes, recovery metrics, therapeutic efficacy, inflammatory markers, and safety profiles to provide evidence for clinical decision-making.

ELIGIBILITY:
Inclusion Criteria:

* Patients who met the diagnostic criteria for acute cholangitis according to the Tokyo Guidelines 2018 (TG18), and were diagnosed through physical examination, ultrasound, CT, or MRCP showing common bile duct stones as the cause of obstruction.
* Body temperature <36°C or >38°C.
* Presence of jaundice or signs of organ dysfunction (e.g., hypotension responsive to fluids for Grade II, or requiring vasopressors for Grade III, altered mental status, etc.).
* Patients who signed informed consent.

Exclusion Criteria:

* Patients with concurrent diseases such as gastric perforation or active gastrointestinal bleeding unrelated to cholangitis.
* Patients with acute pancreatitis as the primary diagnosis.
* Patients with serious primary diseases in the heart, brain, lungs, kidneys, hematopoietic, or nervous systems contraindicating either procedure.
* Pregnant or breastfeeding women.
* Patients with cognitive dysfunction unable to provide consent.
* Known pancreatobiliary malignancy as the cause of obstruction.
* Severe liver cirrhosis (Child-Pugh C) or liver atrophy.
* Patients with severe systemic primary diseases, who could not tolerate the anesthesia or procedure.
* Patients with mental disorders, hematologic diseases (e.g., severe coagulopathy uncorrectable pre-procedure), autoimmune diseases directly impacting biliary system, or those using high-dose corticosteroids affecting inflammatory markers.
* Patients participating in other clinical drug trials.
* Previous ERCP or PTBD for the current episode of cholangitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Length of Hospital Stay | At hospital discharge (up to approximately 3-4 weeks post-procedure).
  The total number of days from hospital admission to discharge.

SECONDARY OUTCOMES:
Time to First Ambulation | From date of procedure until hospital discharge (estimated maximum of 4 weeks).
  Time in days from the procedure until the patient is first able to walk.
Procedure Time | Measured intraoperatively
  Time in minutes from scope insertion/skin puncture to the end of drainage placement.
Time to Return of Bowel Function | From date of procedure until hospital discharge (estimated maximum of 4 weeks).
  Time in hours or days from the procedure until the first flatus or bowel movement.
Change in Inflammatory Markers | Baseline (pre-treatment), 72 hours post-procedure, and 3 months post-treatment.
  Change from baseline in serum levels of Interleukin-6 (IL-6), Interleukin-1 (IL-1), Tumor Necrosis Factor-alpha (TNF-α), and C-reactive protein (CRP).
Change in Pain Intensity | Baseline (pre-treatment), 72 hours post-procedure, and 3 months post-treatment.
  Change from baseline in pain severity assessed using the Visual Analog Scale (VAS), scored 0-10.
Therapeutic Efficacy | Assessed at 24 hours post-procedure.
  Assessed as Significant Effect, Effective, or Ineffective based on resolution of biliary obstruction and clinical symptoms within 24 hours. The total effective rate is calculated as (Significant + Effective) / Total cases.
Incidence of Complications | up to 3 months post-procedure.
  Number of participants experiencing adverse events, including post-ERCP pancreatitis, abdominal infection, gastrointestinal bleeding, bile leakage, liver damage, and procedure-specific complications.

CONTACTS AND LOCATIONS:
Locations (1):
- Wuhan No.1 Hospital (Wuhan Hospital of Traditional Chinese & Western Medicine), Wuhan, Hubei, China